CLINICAL TRIAL: NCT02931617
Title: Comparison of Two Modes of Respiratory Physiotherapy in Cardio-thoracic Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETLR13037
Record Dates: First submitted 2015-12-09; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery; Postoperative; Dysfunction Following Lung Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy w/Positive end expiratory pressure training (Active Comparator): Chest Physiotherapy w/Positive end expiratory pressure training; post therapy lung volume measurements
  Interventions: Other: Chest Physiotherapy; Device: Post-therapy lung volume measurements
- Physiotherapy w/Inspiratory force training (Experimental): Chest Physiotherapy w/Inspiratory force training; post therapy lung volume measurements
  Interventions: Other: Chest Physiotherapy; Device: Post-therapy lung volume measurements

INTERVENTIONS:
Other: Chest Physiotherapy
Device: Post-therapy lung volume measurements — In both intervention groups.

SUMMARY:
Two forms of pre and postoperative physiotherapy are compared in three cohorts of patients undergoing cardio-thoracic surgery: Minor thoracic surgery (biopsy), major thoracic surgery (lobectomy etc, open or VATS) and cardiac surgery

DETAILED DESCRIPTION:
Inspiratory force calibrated training is applied in a controlled randomized trial

ELIGIBILITY:
Inclusion Criteria:

* cardiothoracic operation,
* informed consent

Exclusion Criteria:

* reduced co-operation (such as psychiatric diagnosis),
* severe neurologic disease affecting respiratory function,
* alcohol or drug abuse at hospital entry,
* tuberculosis or other contagious lung infection,
* severe respiratory insufficiency SpO2 < 90 or blood pO2 <8 or rep.rate > 25/min at rest or supplementary oxygen required at home,
* cardiac pacemaker.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 | Preop + 1-3 postoperative days
  Serial measurements
Number of patients with atelectasis | Preop + 1-3 postoperative days
  In chest x-ray
Change in peripheral oxygen saturation | Preop + 1-3 postoperative days
  Serial measurements
Postoperative lung complications | Preop + 1-30 postoperative days
  Number of patients with lung infections, prolonged air leak, pneumothorax

SECONDARY OUTCOMES:
Compliance to Chest physiotherapy | Preop + 1-3 postoperative days
  Serial evaluations and measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jari O Laurikka, MD,PhD, Principal Investigator — Tampere Univeristy Hospital
Locations (1):
- Tampere University Hospital, Heart Center, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lahteenmaki S, Juutinen M, Viik J, Mahrberg H, Laurikka J. Effects of physiotherapy on breathing cycle after thoracic surgery measured with impedance pneumography in a prospective clinical comparison. Gen Thorac Cardiovasc Surg. 2025 Sep 26. doi: 10.1007/s11748-025-02199-y. Online ahead of print. PMID 41004114